CLINICAL TRIAL: NCT02095392
Title: The Effect of Soluble Phosphate in Combination With Different Calcium Doses on Calcium and Phosphorus Metabolism in Healthy Adults
Brief Title: Effects of Soluble Phosphate in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Glei, Prof. Dr., University of Jena
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H55-14
Record Dates: First submitted 2014-03-17; First posted 2014-03-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers
Keywords: soluble phosphate; phosphorus metabolism; calcium metabolism; bone metabolism; human study
MeSH Terms: interventions — Flavonoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- P1000/Ca0 (Experimental)
  Interventions: Dietary Supplement: P1000/Ca0; Dietary Supplement: Placebo
- P1000/Ca500 (Experimental)
  Interventions: Dietary Supplement: P1000/Ca500; Dietary Supplement: Placebo
- P1000/Ca1000 (Experimental)
  Interventions: Dietary Supplement: P1000/Ca1000; Dietary Supplement: Placebo
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: P1000/Ca0; Dietary Supplement: P1000/Ca500; Dietary Supplement: P1000/Ca1000

INTERVENTIONS:
Dietary Supplement: P1000/Ca0 — 22 subjects consume for 8 weeks a beverage enriched with phosphate [1g phosphorus/d]
  Arms: P1000/Ca0; Placebo
Dietary Supplement: P1000/Ca500 — 22 subjects consume for 8 weeks a beverage enriched with phosphate [1 g phosphorus/d] and calcium [0,5 g calcium]
  Arms: P1000/Ca500; Placebo
Dietary Supplement: P1000/Ca1000 — 22 subjects consume for 8 weeks a beverage enriched with phosphate [1 g phosphorus/d] and calcium [1 g calcium]
  Arms: P1000/Ca1000; Placebo
Dietary Supplement: Placebo — all participants consume two weeks before intervention the beverage without phosphate and calcium
  Arms: P1000/Ca0; P1000/Ca1000; P1000/Ca500

SUMMARY:
The study was conducted to investigate the effect of soluble phosphate in combination with different calcium doses on calcium and phosphorus metabolism and further physiological parameters in healthy subjects. The main aim of the study is to investigate the influence of a soluble phosphate supplementation on the fasting blood phosphate concentration and the dependency of an additional calcium intake.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-60 years
* physical health

Exclusion Criteria:

* postmenopausal women
* kidney diseases
* diabetes mellitus
* metabolic diseases
* osteoporosis
* intake of dietary supplements
* pregnancy and lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Fasting phosphate concentration in blood | 8 weeks

SECONDARY OUTCOMES:
Calcium and phosphorus metabolism | 8 weeks
  * parameters of phosphate and calcium metabolism (1,25-OHD; 25-OHD;FGF23;PTH)
  * parameters of bone formation and resorption (osteocalcin, P1NP, CTX)
  * minerals in plasma, faeces and urine

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glei, Prof. Dr., Principal Investigator — Friedrich-Schiller-University Jena, Institute of Nutrition, Department of Nutritional Toxicology
Locations (1):
- Friedrich-Schiller-University Jena, Institute of Nutrition, Department of Nutritional Toxicology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Trautvetter U, Camarinha-Silva A, Jahreis G, Lorkowski S, Glei M. High phosphorus intake and gut-related parameters - results of a randomized placebo-controlled human intervention study. Nutr J. 2018 Feb 16;17(1):23. doi: 10.1186/s12937-018-0331-4. PMID 29452584
- [Derived] Trautvetter U, Jahreis G, Kiehntopf M, Glei M. Consequences of a high phosphorus intake on mineral metabolism and bone remodeling in dependence of calcium intake in healthy subjects - a randomized placebo-controlled human intervention study. Nutr J. 2016 Jan 19;15:7. doi: 10.1186/s12937-016-0125-5. PMID 26786148